CLINICAL TRIAL: NCT02232230
Title: A Multicenter Trial Enrolling Men With Advanced Prostate Cancer Who Are to Receive Combination Radiation and Sipuleucel-T
Status: Completed | Type: Observational
Sponsor: GenesisCare USA (Other)
Collaborators: Dendreon (Industry)
Responsible Party: Sponsor
Other Study IDs: 21C-2013-02
Record Dates: First submitted 2014-07-18; First posted 2014-09-05 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Castrate Refractory Metastatic Prostate Cancer (mCRPC)
MeSH Terms: interventions — sipuleucel-T

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Provenge

SUMMARY:
Radiation in combination with Provenge based immunotherapy may improve outcomes seen on imaging as well as immunologic monitoring. This study will assess the effect of radiation therapy to augment anti-tumor responses from immune therapy with Provenge.

DETAILED DESCRIPTION:
It is common knowledge that the host can make anti-tumor immune responses, although often these are ineffective in causing tumor regression. Boosting these responses with immunotherapy is therefore an attractive, relatively benign adjunctive cancer treatment. Little is known in regards to how standard anti-cancer therapies like radiation therapy might interact with immunotherapy in a clinical setting. We are interested in knowing if the tumor cell death occasioned by radiation therapy might augment anti-tumor responses from the immune therapy, Provenge.

The tentative assumption is that cell death following radiation therapy will stimulate anti-tumor immunity, which could provide a more permanent solution to curing cancer and discouraging tumors from spreading throughout the body. In order to find out if this assumption is correct, for patients undergoing radiation 28 days prior to Provenge, highly developed, laboratory analyses for tumor-specific immunity and imaging will be performed.

ELIGIBILITY:
Inclusion Criteria: Subjects will be recruited from the population of patients who are castrate refractory metastatic prostate cancer (mCRPC) and have made the decision to be treated with radiation therapy to one or more metastatic sites of concern followed at least 28 days later by Provenge.

Exclusion Criteria: The potential subject is unwilling or hesitant to participate for any reason and/or fails to complete the appropriate Informed Consent Form.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with castrate refractory metastatic prostate cancer (mCRPC).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Change in immune stimulation | At 52 Weeks post first injection of sipuleucel-T
  The percentage of subjects who exhibit a two-fold increase in peripheral immune response at any post-treatment time point (6, 10, 14, 26, 39 and 52 weeks after the first infusion of sipuleucel-T) utilizing IFNγ ELISPOT response to PA2024.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Finkelstein, MD, Principal Investigator — GenesisCare USA
Locations (1):
- 21st Century Oncology, Scottsdale, Arizona, United States